CLINICAL TRIAL: NCT02036346
Title: The Effect of Ileostomy Formation on Nutritional Status and Electrolyte Profile in Rectosigmoidectomy Patients: a Prospective Randomized Trial.
Brief Title: Electrolyte Profile, Nutritional Status and Ileostomy Formation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Larissa University Hospital (Other)
Collaborators: University of Thessaly (Other)
Responsible Party: Principal Investigator, ATHANASIOS MIGDANIS, SRD, M.Sc., Larissa University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LarissaUH
Record Dates: First submitted 2013-12-30; First posted 2014-01-15 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Colorectal Resection; Ileostomy
Keywords: ileostomy; colorectal resection; dehydration; nutritional status
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Oral rehydration solution (Experimental): Patients who have undergone colorectal resection surgery resulting in an ileostomy creation
  Interventions: Dietary Supplement: Oral Ηydration Solution
- No intervention (Experimental): Patients who have undergone colorectal resection surgery resulting in an ileostomy creation
  Interventions: Other: Advise on calculated oral fluid requirements
- Colorectal resection without an ileostomy (Active Comparator): Patients who have undergone colorectal resection surgery without an ileostomy creation
  Interventions: Other: No nutritional advice will be given

INTERVENTIONS:
Dietary Supplement: Oral Ηydration Solution — Oral rehydration solution containing: sodium chloride, sodium citrate, glucose, magnesium citrate, food additives and water.
  Arms: Oral rehydration solution
Other: Advise on calculated oral fluid requirements
  Arms: No intervention
Other: No nutritional advice will be given
  Arms: Colorectal resection without an ileostomy

SUMMARY:
One of the main reasons for hospital readmission in ileostomy patients is fluid and electrolyte abnormalities. Prospective observational studies have suggested an occurrence rate of around 20%. Due to colonic exclusion ileostomy patients lose large amounts of sodium and fluid through their stoma effluent. In addition studies have shown that ileostomy construction is a risk factor for renal impairment, occurring secondary to dehydration.

Encouraging patients to increase total fluid intake seems to be a common mistake in clinical practice as this can dilute sodium levels even more, causing greater sodium depletion. In terms of addressing the problem a few small studies have used isotonic drinks of various compositions showing increased electrolyte absorption.

Other dietary complications sometimes include hypomagnesaemia and decreased absorption of B-12 and folic acid, however due to the integrity of the small intestine other nutrient malabsorption is unlikely to occur. As far as body composition is concerned obesity has been shown to be a risk factor for peri- and postoperative complications in colorectal surgery (e.g. peristomal dermatitis, stoma stenosis and prolapse). A prospective trial examining measures that can prevent readmission for dehydration and other nutritional considerations related to this group of patients is definitely required.

Hypothesis:

The administration of an oral rehydration solution will allow a significant decrease in dehydration and electrolyte abnormality rates in patients with a temporary ileostomy.

ELIGIBILITY:
Inclusion Criteria:

* Male of female patients of more than 18 years of age
* Patients who have undergone a rectosigmoidectomy procedure resulting or not in an ileostomy formation

Exclusion Criteria:

* Short Bowel Syndrome
* Diabetic ketoacidosis
* Chronic Renal failure
* Hepatic/Cardiac failure
* Diabetes insipidus
* Diuretic Medication
* Corticosteroid Medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2013-12; Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Serum electrolyte levels | up to 20-40 days postoperatively
  sodium (mmol/l)
Serum electrolyte levels | up to 20-40 days postoperatively
  potassium (mmol/l)
Serum electrolyte levels | up to 20-40 days postoperatively
  magnesium (mg/dl)
Serum electrolyte levels | up to 20-40 days postoperatively
  chloride (mmol/l)

SECONDARY OUTCOMES:
Physical findings of dehydration | 20 days postoperatively, 40 days postoperatively
  thirst, dizziness, lethargy, oliguria, dense urine
Biochemical markers reflecting dehydration and renal function | 20 days postoperativey, 40 days postoperatively
  Urea (mg/dl)
Biochemical markers reflecting dehydration and renal function | 20 days postoperativey, 40 days postoperatively
  Creatinine (mg/dl)
Anthropometric characteristics | baseline, 40 days postoperatively
  weight (kg)
Anthropometric characteristics | baseline, 40 days postoperatively
  height (m)
Anthropometric characteristics | baseline, 40 days postoperatively
  BMI (kg/m2)
Anthropometric characteristics | baseline, 40 days postoperatively
  total body fat (%)
Nutritional Intake | baseline, at 20 days and 40 days postoperatively
  Energy intake assessed through 24hour recalls and analyzed via nutrition analysis software
Nutritional Intake | baseline, at 20 days and 40 days postoperatively
  Macronutrient intake assessed through 24hour recalls and analyzed via nutrition analysis software
Nutritional Intake | baseline, at 20 days and 40 days postoperatively
  Electrolyte intake via diet assessed through 24hour recalls and analyzed via nutrition analysis software
Stoma output (ml/L) | baseline, at 20 days and 40 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: GEORGE TZOVARAS, MD, Study Chair — University Hospital of Larissa; GEORGE TZOVARAS, MD, Study Director — University Hopsital of Larissa; Georgios D Koukoulis, M.D. MSc PhD, Principal Investigator — Department of General Surgery, University Hospital of Larisa
Locations (1):
- University Hospital of Larissa, Larissa, Thessaly, Greece

REFERENCES:
- [Background] Migdanis A, Koukoulis G, Mamaloudis I, Baloyiannis I, Migdanis I, Kanaki M, Malissiova E, Tzovaras G. Administration of an Oral Hydration Solution Prevents Electrolyte and Fluid Disturbances and Reduces Readmissions in Patients With a Diverting Ileostomy After Colorectal Surgery: A Prospective, Randomized, Controlled Trial. Dis Colon Rectum. 2018 Jul;61(7):840-846. doi: 10.1097/DCR.0000000000001082. PMID 29771807
- [Derived] Migdanis A, Koukoulis G, Mamaloudis I, Baloyiannis I, Migdanis I, Vagena X, Malissiova E, Tzovaras G. The effect of a diverting ileostomy formation on nutritional status and energy intake of patients undergoing colorectal surgery. Clin Nutr ESPEN. 2020 Dec;40:357-362. doi: 10.1016/j.clnesp.2020.08.002. Epub 2020 Aug 28. PMID 33183563
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/29771807